CLINICAL TRIAL: NCT00628550
Title: A Prospective, Randomized, Controlled Trial of Combination Vasopressin and Epinephrine to Epinephrine Only for In-Intensive Care Unit Pediatric Cardiopulmonary Resuscitation
Brief Title: Trial of Vasopressin and Epinephrine to Epinephrine Only for In-Hospital Pediatric Cardiopulmonary Resuscitation
Acronym: Vasopressin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 082007-065
Record Dates: First submitted 2008-02-24; First posted 2008-03-05 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cardiopulmonary Arrest; Cardiac Arrest
Keywords: cardiac arrest; cardiopulmonary arrest; vasopressin; epinephrine; pediatrics; in hospital cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Diabetes Insipidus | interventions — Vasopressins; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pediatric patients that experience in-hospital CPA who remain in cardiac arrest despite CPR and an initial, standard dose of epinephrine (0.01 mg/kg), will be randomly assigned to receive vasopressin (0.8 units/kg) rescue as the second vasopressor medication.
  Interventions: Drug: Vasopressin
- 2 (Active Comparator): Pediatric patients that experience in-hospital CPA who remain in cardiac arrest despite CPR and an initial, standard dose of epinephrine (0.01 mg/kg), will be randomly assigned to receive standard dose epinephrine (0.01 mg/kg)rescue as the second vasopressor medication.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Vasopressin — One dose of vasopressin (0.8 units/kg) intravenously rescue as the second vasopressor medication.
  Other Names: Pitressin
  Arms: 1
Drug: Epinephrine — One standard dose epinephrine (0.01 mg/kg) intravenously rescue as the second vasopressor medication.
  Other Names: Adrenaline
  Arms: 2

SUMMARY:
Cardiac arrest has a very poor prognosis, especially with prolonged efforts at resuscitation, and unfortunately, survivors are often severely neurologically impaired. CPA in children is often the result of a prolonged illness rather than a sudden, primary cardiac event as is frequent in adults. This necessitates that resuscitation research must be conducted separately for pediatric and adult patients. Authorities currently endorse the use of epinephrine for restoring spontaneous circulation based on its ability to maintain diastolic blood pressure and subsequent blood flow to the heart during resuscitation. However, human studies have shown no clear survival benefit of epinephrine and have elucidated concerning adverse effects. Recently, both the European Resuscitation Council and the American Heart Association have recognized the use of vasopressin as a promising vasoconstrictor and an alternative or adjunct to epinephrine in the resuscitation of adults. Vasopressin causes profound vasoconstriction without the adverse effects of epinephrine and is associated with improved blood flow to the heart and brain. This increased cerebral blood flow has been associated with better neurologic outcome in animal studies. In light of compelling animal and human studies of combined vasopressin and epinephrine, pediatric trials are indicated for vasopressin usage in pediatric CPR. This study will evaluate the addition of the administration of vasopressin to standard advanced CPR therapy (epinephrine alone) for pediatric patients that experience in-intensive care unit CPA to assess for improved time to return of spontaneous circulation (ROSC), survival to 24 hours, survival to hospital discharge, and neurologic outcome. When a patient experiences a CPA, standard Pediatric Advanced Life Saving (PALS) protocols as endorsed by the American Heart Association will be initiated. This will include receiving epinephrine as the first vasopressor medication. Patients will then be randomized to receive vasopressin (treatment group) or epinephrine (control group) as the second vasopressor medication, if needed. If more then two doses of vasopressor medication is required in either group, epinephrine will be administered according to the PALS algorithm until the end of the event. All CPA events meeting inclusion criteria will be entered into the National Registry of Cardiopulmonary Resuscitation (NRCPR) Database, which tracts all CPA events at Children's Medical Center Dallas. Prior to commencement of the RCT, a pilot trial of 10 patients will be completed to assess preliminary safety, feasibility, and effectiveness of combination epinephrine-vasopressin for pediatric in-intensive care unit CPA refractory to initial epinephrine dosing. All pilot patients will receive vasopressin as the second vasopressor medication.

DETAILED DESCRIPTION:
CONCISE SUMMARY OF PROJECT:

The study design will be a prospective, randomized, controlled clinical trial to be conducted in the PICU of CMC Dallas (UT Southwestern Medical Center) following a pilot trial enrolling 10 patients. This study will be undertaken after consultation with and acceptance by the resuscitation committee and PICU at CMC. Pediatric patients that experience in-hospital CPA who remain in cardiac arrest despite CPR and an initial, standard dose of epinephrine (0.01 mg/kg), will be randomly assigned to receive either standard dose epinephrine (0.01 mg/kg) or vasopressin (0.8 units/kg) rescue as the second vasopressor medication.

SUMMARY OF STUDY PROCEDURES:

When a patient experiences a CPA, standard Pediatric Advanced Life Saving (PALS) protocols will be followed. This will include: establishment of an airway, support of breathing including supplemental oxygen, evaluation of cardiac rhythm, chest compressions, electrical defibrillation if appropriate, and administration of epinephrine as the first vasopressor medication. The quality of CPR will be monitored and reported by the documenting nurse for the event, to include rate of ventilation, rate and depth of chest compressions, and no-flow time (time without chest compressions). In addition, monitoring of end-tidal CO2, diastolic blood pressure via arterial line if present, and human observation and coaching will be employed to track CPR quality. The patient will then be randomized to receive either epinephrine (control group) or vasopressin (treatment group) as the second vasopressor medication if needed. If further doses of medication are required in either group, epinephrine will be administered according to the PALS algorithm until the end of the CPA event as defined below. Thus, the only difference between the groups will be the replacement of epinephrine with vasopressin as the second vasopressor medication in the algorithm. A total of 120 patients will be enrolled in the randomized, controlled trial portion of the study.

After completion of PICU staff training and prior to the randomized, controlled trial, a pilot trial of vasopressin resuscitation involving 10 patients will be conducted to test the feasibility and safety of study methodology. Pilot participants who meet inclusion criteria will be enrolled serially from the PICU at CMC. Study protocol for the treatment group of the randomized, control trial (vasopressin + epinephrine) will be followed. Collected information will be reviewed by members of a Data Safety and Monitoring Board (DSMB) before proceeding to the next phase of the trial. These patients will not be included in the final analysis.

The requirement of two doses of resuscitation medications will provide adequate time for randomization and use of vasopressin. It will also exclude those children with rapidly reversible conditions who would not have time to benefit from vasopressin versus epinephrine intervention. Stratified randomization technique will be used to control for the effect of vasopressor infusions the patient is receiving at the time of cardiac arrest. Stratification will be based on 4 groups i.e., epinephrine, vasopressin, both, or neither. In order to avoid extreme imbalance in the size of the treatment arms, a permuted block design will be used and the size of each block will be set at 6. SPSS pseudo-random number generator will be used to design the randomization charts. Randomization will be accomplished by the PICU pharmacist via sealed envelopes designating study arm assignment that will be available on every code cart in the PICU. Thus, the study medication will be blinded to all but the pharmacist.

On admission to the PICU, families of all patients will be informed and educated of this ongoing study with exception from informed consent (EFIC) via posters in the waiting rooms and a brochure regarding the study clearly explaining how to "opt out" of inclusion. The number of patients who "opt out" of inclusion will be documented and available to the IRB at their request. Representatives of the study will be available by phone 24 hours a day and in person in the waiting room daily to discuss the study and answer questions. Parents will be informed of inclusion within 24 hours in person or by phone or letter if unavailable. This notification will be documented and consent will be elicited for follow up data collection. CPA events will be limited to those occurring in the PICU only. Providers that respond to CPA events will be in-serviced regarding the study protocol prior to implementation via didactic sessions. Input from pharmacists and providers in the PICU will be sought to assure the easiest implementation possible. Vasopressin is currently available for administration on all resuscitation (code) carts at CMC. Inclusion and exclusion criteria will be posted on all code carts to assist providers. Current protocol at CMC to enter all CPA events into the National Registry of Cardiopulmonary Resuscitation (NRCPR) will be followed. This data is a complete account of the events of the CPA and will be sufficient to meet all of the study's stated goals and objectives. Only data pertinent to the outcomes of this study will be reviewed from the database. This data will also be reviewed to assure standardization of execution of the study protocol.

Time to Completion Given that 89 CPA events met inclusion criteria from January 2005 to June 2006 in the PICU at CMC, approximately 30 months will be required to enroll 130 total patients into this study (10 patients in pilot trial, 120 patients in main study). Subjects will be enrolled in the study until discharge or in-hospital death.

Definition CPA End of Event

1. . ROSC that is sustained for > 20mins with no further need for chest compressions, including with a pacemaker or extracorporeal membrane oxygenation OR
2. . Resuscitation event is terminated and patient is declared dead (unresponsive to advanced life support, medical futility, advance directive, restriction by family member)

SPECIAL PRECAUTIONS:

A full resuscitation team will be present whenever vasopressin is administered including a physician, nurse, respiratory technician, clinical technician, and pharmacist. A sign will be clearly posted on the bed of any patient whose proxy has "opted" the patient out of the study or who meets any other exclusion criteria. The DSMB will evaluate the study for clear benefit or harm, lack of efficacy, or unacceptable toxicity of vasopressin.

SOURCES OF RESEARCH MATERIALS/ COLLECTION OF FOLLOW UP DATA:

Data from CPA events will be collected from the NRCPR database which is completed at the conclusion of every CPA event currently at CMC. Data is collected in six major categories of variables: (1) Facility data, (2) Patient demographic data, (3) Pre-event data, (4) Event data, (5) Outcome data, and (6) Quality improvement data. All patient identifiers will be destroyed at the earliest possible opportunity. Data will be de-identified for analysis. This data will include laboratory and treatment data from the hospitalization in the PICU at CMC before, during, and after resuscitation. Specifically, this data will include: age, gender, vital signs, treatments, laboratory results, neurologic exam (PCPC and POPC scores) and physical exam. The data collection is based on in-hospital Utstein-style guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All children, ages 0 to 18 years, admitted to the PICU who experience CPA requiring either chest compressions and/or defibrillation. This will include males, females and Spanish speaking individuals.
* Patients must require at least 2 doses of vasopressor medication during the CPA event (all patients would receive epinephrine as first dose, followed by either epinephrine or vasopressin as second dose depending on randomization, all subsequent doses required would be epinephrine) given via any route (intravenous, intraosseous, or endotracheal).

Exclusion Criteria:

* Do Not Attempt Resuscitate (DNAR) patients
* Chemical code only (i.e., no CPR/defibrillation)
* Events not requiring chest compressions and/or defibrillation
* Events with a pulse requiring synchronized or unsynchronized cardioversion
* Successful internal cardiac device defibrillation of Vfib/pVT that initiates the resuscitation event
* Defibrillation for Vfib/pVT without administration of a vasopressor
* All patients in the custody of the State of Texas
* Any patient whose parent or guardian "opts out" of the study
* Any patient who is pregnant
* Any patient whose attending physician "opts out" of the study
* Any patient who does not consent to follow up data collection

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Combination vasopressin and epinephrine (CPA refractory to cardiopulmonary resuscitation and initial epinephrine dosing) will increase the proportion of patients surviving to hospital discharge by 25% compared to epinephrine alone. | Immediate

SECONDARY OUTCOMES:
Combination vasopressin and epinephrine will decrease the time to ROSC | Immediate
Vasopressin and epinephrine will improve the proportion of CPA survivors with favorable neurologic outcome (short-term Pediatric Overall Performance Category) [POPC] score discharge of 1-3 or unchanged from hospital admission at the time of hospital . | Period of hospitalization
Vasopressin and epinephrine will improve the proportion of CPA survivors with favorable neurologic outcome (short-term Pediatric Cerebral Performance Category) [PCPC] score of 1-3 or unchanged from hospital admission at time of hospital discharge. | Period of Hospitalization
Combination vasopressin and epinephrine will improve 24 hour survival. | 24 hrs
Combination vasopressin and epinephrine will decrease the proportion of patients who require prolonged CPR (CPR > 20minutes) to achieve sustained ROSC. | Immediate
Combination vasopressin and epinephrine will increase organ recovery in those patients who meet brain death criteria following the CPA event. | Period of hospitalization
Combination epinephrine and vasopressin will improve rates of return of spontaneous circulation (ROSC) | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Tia Tortoriello Raymond, M.D., Principal Investigator — Universtiy of Texas Southwestern
Locations (1):
- Universtity of Texas Southwestern, Children's Medical Center, Dallas, Texas, United States